CLINICAL TRIAL: NCT02241109
Title: Predicting Aortic Stenosis Progression by Measuring Serum Calcification Propensity
Acronym: PASP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 087/14
Record Dates: First submitted 2014-09-11; First posted 2014-09-16 (Estimated); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Aortic Valve Sclerosis; Aortic Valve Stenosis; Stenosis Progression; Valvular Heart Disease
Keywords: aortic stenosis progression; aortic valve sclerosis progression; calcification propensity
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients (Other): Compare patients with high calcification propensity do have faster valve-stenosis progression
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — progression monitoring by echocardiography

SUMMARY:
Aortic stenosis is the most common valvular heart disease and an important public-health problem. Surgical or interventional aortic valve replacement are based on symptoms and measures of valvular and ventricular function using echocardiography.There is no uniform pattern of progression. Instead, marked differences not only between individuals, but also during the time course of the disease can be observed.

Several prospective studies have been performed to enhance the predictability of disease behavior. Individually it is still prone to large errors and hard to predict aortic stenosis progression. Therefore, in patients with aortic sclerosis without severe stenosis, it is desirable to find a strong predictor of rapid disease progression. This would allow anticipating cardiovascular deterioration by identifying individuals at particular risk.

Study Hypothesis

In patients with aortic sclerosis, increased serum calcification propensity, as measured by the T50-Test, is related to the amount of stenosis progression in one year.

DETAILED DESCRIPTION:
Background

Clinical Background

Aortic stenosis is the most common valvular heart disease and an important public-health problem. It is present in approximately 25% of all adults aged >65 years. Decisions about surgical or interventional aortic valve replacement are based on symptoms and measures of valvular and ventricular function using echocardiography. Such valvular affections are the result of a chronic progressive disease, usually starting with hemodynamically non-significant aortic sclerosis, and then progressing to severe stenosis over years. There is no uniform pattern of progression. Instead, marked differences not only between individuals, but also during the time course of the disease can be observed. Aortic sclerosis progresses to mild aortic stenosis in <15% of patients over 2 to 7 years. Once moderate stenosis is present (jet velocity >3 m/s), the average progression is 0.3 m/s per year, but still highly variable. When peak jet velocity exceeds 4 m/s, survival free from symptoms and valve replacement is significantly reduced.

In the past, several prospective studies have been performed to enhance the predictability of disease behavior. Some determinants of rapid progression and adverse outcome have been identified, such as: age, gender, cardiovascular risk factors, B-natriuretic peptide, stenosis severity, degree of valvular calcification and others. Although it appears that progression is more rapid in degenerative calcific disease than congenital or rheumatic disease, predicting progression individually is still prone to large errors even when considering these determinants. Therefore, regular clinical follow-up is mandatory in patients with asymptomatic aortic valve affections. In patients with aortic sclerosis without severe stenosis, it is desirable to find a strong predictor of rapid disease progression. This would allow anticipating cardiovascular deterioration by identifying individuals at particular risk.

Background of Tissue Calcification

From a biochemical and histological point of view, aortic sclerosis is a valvular disease characterized by focal plaque-like lesions containing microscopic calcifications. Because calcium and phosphate concentrations in serum are near supersaturation, the balance of inhibitors and promoters critically influences the development of calcification. The serum protein fetuin-A is a major systemic inhibitor of calcification. Together with additional blood components, fetuin-A prevents the supersaturated calcium and phosphate from precipitating by forming soluble colloidal protein-mineral nanoparticles and is therefore an integral part of the defense system preventing calcifications. Low serum concentrations of fetuin-A are associated with a reduced capacity to inhibit calcification in vitro. Calcification takes place when this humoral line of defense is overwhelmed.

Koos et al. showed that serum levels of the calcification inhibitor fetuin-A are associated with the progression of aortic valve calcifications and major adverse clinical events, independent of the renal function and inflammation.

A novel in vitro blood test developed by Pasch et al. provides an overall measure of calcification propensity by monitoring the maturation time (T50) of calciprotein particles. First published clinical data indicate that the T50 test is a helpful biomarker for the prediction of future vascular calcifications.

Study Endpoints

* Index test (parameter to be evaluated): T50-Test
* Comparator tests (tests to define disease status):

Primary:

Progression of peak aortic jet velocity over one year (m/s per year)

Secondary:

Progression of peak aortic jet velocity >20% in one year (dichotomized primary comparator) Combined endpoint: death, hospitalizations, aortic-valve replacement, heart failure, angina, syncope

Inclusion Criteria

* Patient referred to routine clinical echocardiography at the Department of Cardiology, Inselspital Bern
* Aortic sclerosis with or without stenosis
* Written informed consent

Exclusion Criteria

The goal is to recruit a population comprising a large variety of clinical conditions. Exclusion criteria are:

* Age <18 years
* Aortic valve replacement scheduled within 1 year after inclusion
* Any aortic valvular disease other than degenerative sclerotic, bi- or unicuspid valves
* Known disease with expected survival <1 year
* Known malignant tumor
* Subvalvular obstruction (in LVOT) with mean pressure gradient >10mmHg

Echocardiography

Patients will be examined by standard echocardiography including a comprehensive assessment of cavity and wall dimensions, ventricular and valvular function, morphologic appraisal and pressure predictions. In particular, peak aortic jet velocity will be recorded using CW Doppler from the window yielding the highest velocity signal. Aortic stenosis severity will be measured using peak flow velocity (m/s). Progression will be expressed as peak flow velocity change per year (m/s per year). Aortic valve sclerosis will be assessed visually from a short axis according to Rosenhek: 1, no calcification; 2, mildly calcified (small isolated spots); 3, moderately calcified (multiple larger spots); and 4, heavily calcified (extensive thickening and calcification of all cusps).

T50-Test The addition of calcium and phosphate to serum triggers the formation of primary calciprotein particles (CPP, see figures 2 and 3). As nano-suspension of calcium-phosphate, these particles represent a defense mechanism of the serum against calcification. Primary CPPs undergo spontaneous transition to secondary CPPs. The formation of these particles represents calcification. In the T50-Test, the time elapsed for the transformation of 50% of the particles is measured and is specific for individual sera.

The blood-sample will be taken immediately after completion of the echocardiographic exam.

Objective

The purpose of this study in patients with aortic sclerosis with and without stenosis is to establish an independent predictor of progression of aortic valve obstruction using a new calcification propensity measure in the serum.

Methods

Recruitment 200 consecutive patients referred for a routine clinical echocardiographic exam showing varying degrees of aortic sclerosis will be included.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred to routine clinical echocardiography
* Aortic sclerosis with or without stenosis
* Written informed consent

Exclusion Criteria

* Age <18 years
* Aortic valve replacement scheduled within 1 year after inclusion
* Any aortic valvular disease other than degenerative sclerotic, bi- or unicuspid valves
* Known disease with expected survival <1 year
* Known malignant tumor
* Subvalvular obstruction (in left ventricular outflow tract) with mean pressure gradient >10mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Progression of peak aortic jet velocity over one year (m/s per year) | One year

SECONDARY OUTCOMES:
Progression of peak aortic jet velocity >20% in one year | One year
Combined endpoint: death, hospitalizations, aortic-valve replacement, heart failure, angina, syncope | One year

CONTACTS AND LOCATIONS:
Overall Officials: Stefano de Marchi, Senior Consultant, Principal Investigator — Dept. of Cardiology, University Hospital Bern, Switzerland
Locations (1):
- Dep. of Cardiology, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Otto CM, Lind BK, Kitzman DW, Gersh BJ, Siscovick DS. Association of aortic-valve sclerosis with cardiovascular mortality and morbidity in the elderly. N Engl J Med. 1999 Jul 15;341(3):142-7. doi: 10.1056/NEJM199907153410302. PMID 10403851
- [Background] Manning WJ. Asymptomatic aortic stenosis in the elderly: a clinical review. JAMA. 2013 Oct 9;310(14):1490-7. doi: 10.1001/jama.2013.279194. PMID 24104373
- [Background] Freeman RV, Otto CM. Spectrum of calcific aortic valve disease: pathogenesis, disease progression, and treatment strategies. Circulation. 2005 Jun 21;111(24):3316-26. doi: 10.1161/CIRCULATIONAHA.104.486738. No abstract available. PMID 15967862
- [Background] Otto CM, Burwash IG, Legget ME, Munt BI, Fujioka M, Healy NL, Kraft CD, Miyake-Hull CY, Schwaegler RG. Prospective study of asymptomatic valvular aortic stenosis. Clinical, echocardiographic, and exercise predictors of outcome. Circulation. 1997 May 6;95(9):2262-70. doi: 10.1161/01.cir.95.9.2262. PMID 9142003
- [Background] Koos R, Brandenburg V, Mahnken AH, Muhlenbruch G, Stanzel S, Gunther RW, Floege J, Jahnen-Dechent W, Kelm M, Kuhl HP. Association of fetuin-A levels with the progression of aortic valve calcification in non-dialyzed patients. Eur Heart J. 2009 Aug;30(16):2054-61. doi: 10.1093/eurheartj/ehp158. Epub 2009 May 8. PMID 19429630
- [Background] Pasch A, Farese S, Graber S, Wald J, Richtering W, Floege J, Jahnen-Dechent W. Nanoparticle-based test measures overall propensity for calcification in serum. J Am Soc Nephrol. 2012 Oct;23(10):1744-52. doi: 10.1681/ASN.2012030240. Epub 2012 Sep 6. PMID 22956818
- [Background] Smith ER, Ford ML, Tomlinson LA, Bodenham E, McMahon LP, Farese S, Rajkumar C, Holt SG, Pasch A. Serum calcification propensity predicts all-cause mortality in predialysis CKD. J Am Soc Nephrol. 2014 Feb;25(2):339-48. doi: 10.1681/ASN.2013060635. Epub 2013 Oct 31. PMID 24179171
- [Background] Rosenhek R, Klaar U, Schemper M, Scholten C, Heger M, Gabriel H, Binder T, Maurer G, Baumgartner H. Mild and moderate aortic stenosis. Natural history and risk stratification by echocardiography. Eur Heart J. 2004 Feb;25(3):199-205. doi: 10.1016/j.ehj.2003.12.002. PMID 14972419